CLINICAL TRIAL: NCT05224323
Title: Avalanche Phenomenon During Airways Opening in Acute Respiratory Distress Syndrome
Acronym: AVALANCHE
Status: Recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AVALANCHE
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Airway pressure, flow, esophageal pressure, ventilation distribution — After informed consent, baseline characteristics of patients will be collected. Airway pressure, flow and esophageal pressure will be recorded using high sampling rate and ventilation distribution using electrical impedance tomography will be recorded during the study. The ventilator will be set at a positive end-expiratory pressure of 15 cmH2O during 10 minutes. Then, respiratory rate will be decreased to 8 breaths/min, and positive end-expiratory pressure will be decreased to 5 cmH2O over one breath to measure the recruited volume. Then, three low-flow inflation and deflation pressure-volume curves will be performed before resuming clinical ventilator settings. Patients will be followed until Day 28 after inclusion or ICU discharge. Maneuvers performed are part of the usual care of patients with acute respiratory distress syndrome in our unit.

SUMMARY:
Acute respiratory distress syndrome accounts for 23% of mechanically ventilated patients and is associated with high mortality rate. Although life-saving, mechanical ventilation may worsen lung injury through two main mechanisms: lung overdistension and atelectrauma. Indeed, the cyclic opening and closure of airways during tidal ventilation may cause lung and bronchial injuries as suggested by animal models and autopsy findings. Complete airways closure has recently been described in 40% of patients with acute respiratory distress syndrome, and setting positive end-expiratory pressure above the airway opening pressure may limit atelectrauma. However, animal and mathematical models suggest that above the airway opening pressure, more distal airways open unevenly according to their own opening pressure, resulting in an "avalanche"-like phenomenon during lung inflation. This phenomenon has never been described in humans. A better understanding of the opening of airways in acute respiratory distress syndrome may help to limit ventilation-induced lung injury and to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Moderate-to-severe acute respiratory distress syndrome within the first 72 hours after meeting the Berlin definition criteria:
* Within 1 week of a known clinical insult or new or worsening respiratory symptoms;
* Bilateral opacities (not fully explained by effusions, lobar/lung collapse, or nodules);
* Respiratory failure not fully explained by cardiac failure or fluid overload;
* PaO2/FiO2 ≤ 200 mmHg with positive end-expiratory pressure ≥ 5 cmH2O.
* Absence of spontaneous breathing efforts
* Consent to participate to the study from the patient and/or its surrogate

Exclusion Criteria:

* Pneumothorax
* Broncho-pleural fistula
* Tracheostomy
* Hemodynamic instability
* Severe hypoxemia
* Suspected of proven intracranial hypertension
* Chronic obstructive lung disease
* Pacemaker or defibrillator
* Decision to withhold of withdraw life-sustaining measures
* Under protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-to-severe acute respiratory distress syndrome will be included within the first 72 hours after meeting the Berlin definition criteria.
  After ruling out exclusion criteria and obtaining informed consent from their relatives, patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of "avalanche" phenomenon during low-flow lung inflation. | At inclusion
  The distribution of pressure drops on low-flow inflation pressure-volume curves will be described and plotted on a log-log scale graph. "Avalanche" phenomenon will be defined if this distribution follows power law (i.e. is linear on a log-log scale) with a R2 ≥ 0.80. The prevalence of "avalanche" phenomenon will be described as frequency and 95% confidence interval.

SECONDARY OUTCOMES:
To compare characteristics of patients and their outcomes according to the existence of "avalanche" phenomenon during low-flow lung inflation. | Day 28
  Continuous variables will be summarized as mean ± standard deviation or median [25th-75th percentile] according to their distribution and compared by means of the Mann-Whitney or the Student's t test. Categorical variables will be summarized as frequency (percentage) and 95% confidence interval, and compared by means of Fisher or Chi2 test.
To assess the existence of an inflection point on the low-flow deflation pressure-volume curve. | At inclusion
  The slope of the low-flow deflation pressure-volume curve will be computed by means of linear regression and summarized as mean ± standard deviation or median [25th-75th percentile] according to its distribution. The existence of an inflexion point will be summarized as number (percentage) and 95% confidence interval. The airway pressure corresponding to this inflexion point will be summarized as mean ± standard deviation or median [25th-75th percentile] according to its distribution.
To assess the airway pressure value of the inflection point on the low-flow deflation pressure-volume curve in patients with an inflexion point on the low-flow deflation pressure-volume curve | At inclusion
  The airway pressure corresponding to the inflexion point on the low-flow deflation pressure-volume curve will be summarized as mean ± standard deviation or median [25th-75th percentile] according to its distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suki B, Barabasi AL, Hantos Z, Petak F, Stanley HE. Avalanches and power-law behaviour in lung inflation. Nature. 1994 Apr 14;368(6472):615-8. doi: 10.1038/368615a0. PMID 8145846
- [Background] Chen L, Del Sorbo L, Grieco DL, Shklar O, Junhasavasdikul D, Telias I, Fan E, Brochard L. Airway Closure in Acute Respiratory Distress Syndrome: An Underestimated and Misinterpreted Phenomenon. Am J Respir Crit Care Med. 2018 Jan 1;197(1):132-136. doi: 10.1164/rccm.201702-0388LE. No abstract available. PMID 28557528